CLINICAL TRIAL: NCT07136506
Title: Gait Analysis Parameter and Upper Limb Evaluation in Control Participants
Acronym: ActiControl
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other); SYSNAV (Industry)
Responsible Party: Principal Investigator, Laurent Servais, Principal Investigator, Pediatrician, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ActiControl
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Healthy Volunteers; Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Experimental)
  Interventions: Device: Syde; Other: Post-recording questionnaire

INTERVENTIONS:
Device: Syde — Syde is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.
Other: Post-recording questionnaire — The post-recording questionnaire aims at describing as much as possible the subject activity and quality of life during the recording period while being as low a burden as possible for the subject. The question formats are, on one hand, inspired by Quality of life and Physical Activity questionnaires usually used in Clinical Research and, on the other hand, based on device-specific needs for an optimal analysis. It covers fatigue status, physical status, physical activity with the Syde®, event(s) or condition(s) that may have impacted the ability to wear the Syde® during the recording.

SUMMARY:
The ActiControl study is a monocentric, academic, and fully remote observational study designed to build a normative, longitudinal dataset using the Syde® wearable device. The study will enroll 200 healthy volunteers across all age groups, genders, and backgrounds. Participants will be remotely recruited and followed over two years, wearing the Syde® device for 3-week periods every 6 months. All study visits, including consent, data collection, and follow-up, are conducted remotely via phone or video conferencing. The primary objectives are to collect reference data on gait and movement patterns and to assess adherence and acceptability of the device. Secondary objectives include evaluating the reliability of digital endpoints and the influence of demographic and lifestyle factors on these measures.

DETAILED DESCRIPTION:
Rare diseases, though individually uncommon, collectively affect approximately 5% of the European population, with many presenting neurological symptoms and significant societal burden. Clinical trials in this field face challenges such as small sample sizes and subjective outcome measures. To address these limitations, wearable technologies like Syde® and ActiMyo® have been developed to objectively quantify motor function using inertial sensors.

The Syde® device, worn on the wrist and ankle(s), continuously records upper- and lower-limb movements. One of its key metrics, the 95th percentile of stride velocity (SV95C), has been endorsed by the European Medicines Agency as a valid primary outcome in Duchenne Muscular Dystrophy (DMD) trials. Syde® has also been used in studies involving Spinal Muscular Atrophy (SMA), Angelman Syndrome, Facioscapulohumeral Muscular Dystrophy (FSHD), and other neurological conditions, as well as in healthy controls under 20 years old.

To further validate digital outcome measures, normative data across all age groups is essential. The ActiControl study will enroll 200 healthy volunteers (approximately 20 per decade from ages 0 to 90), ensuring balanced representation by gender, ethnicity, and socioeconomic status.

All study procedures are conducted remotely. Participants are recruited and enrolled electronically, including remote signing of the informed consent form. Demographic and health data (e.g., age, sex, height, weight) are collected via phone or video call at inclusion and every 6 months for 2 years. Participants will wear the Syde® device for 3 weeks at five timepoints (baseline, 6, 12, 18, and 24 months).

Primary objectives include:

Building a longitudinal dataset of Syde® digital variables. Assessing adherence and acceptability of the device across age groups.

Secondary objectives include:

Evaluating the reliability of Syde®-derived variables. Investigating the influence of demographic and lifestyle factors (e.g., age, gender, BMI, physical activity, seasonality) on digital endpoints.

Outcome measures include stride velocity, stride length, walking time, step asymmetry, stair climbing metrics, and more.

This study will contribute to the establishment of robust normative data, enabling more accurate interpretation of digital biomarkers in future clinical trials for rare and neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of different age groups
* Signed informed consent form by participant him/herself or, in case of patients <18 years old, signed informed consent form by patient's parents or legal guardians
* Able to ambulate (minimum 10 meters without help)
* Participants with a reported BMI ≥17 and ≤30
* Participant willing and able to comply with all study procedures

Exclusion Criteria:

* Patients who have undergone a surgical procedure or who have experienced recent trauma (within fewer than 6 months) affecting the upper or lower limbs
* Elite athletes (at the national level)
* Pregnant women
* A chronic or acute muscular, neurological, infectious, or inflammatory pathology within the 3-week period immediately prior to inclusion
* An orthopedic, neuromuscular, or neurological pathology that affects the quality of the participant's walking gait
* No access to unlimited internet connection or alternatively no capacity to come on-site to upload Syde data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Digital Mobility Monitoring Compliance | 5 recording periods of 3 weeks over 2 years
  Measure of participant adherence to wearing the Syde® device using different parameters including total recording time, number of valid recording days (≥4 hours), and time to reach 50 and 180 hours of recording.
Walking Pattern Characteristics | 5 recording periods of 3 weeks over 2 years
  Analysis of walking sequences, including maximal walking sequence duration, maximal distance walked in a single sequence, and maximal 30-minute walking distance.

SECONDARY OUTCOMES:
Device Acceptability and Adherence | 5 recording periods of 3 weeks over 2 years
  Measures of user engagement with the Syde® device across age groups and over time, including total recording time, valid days (≥5 hours), and time to reach 50 and 180 hours.
Reliability of Digital Variables | 5 recording periods of 3 weeks over 2 years
  Test-retest reliability of Syde® digital variables assessed using intraclass correlation coefficients (ICC) between two consecutive half-periods.
Association with Demographic and Health Factors | Over 2 years
  Correlation of digital mobility outcomes with age, height, weight, BMI, and other demographic or health-related variables.
Group Differences in Digital Variables | Over 2 years
  Comparison of digital mobility metrics across subgroups defined by gender, age, health status, education, socio-professional category, physical activity level, living environment, and seasonality.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No